CLINICAL TRIAL: NCT02047747
Title: A Phase II Study to Evaluate the Efficacy, Safety, and Central Nervous System (CNS) Pharmacokinetics of the HER Family Inhibitor Dacomitinib in Progressive Brain Metastases
Brief Title: A Phase II Study of Dacomitinib in Progressive Brain Metastases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow enrollment
Sponsor: David Piccioni, M.D., Ph.D (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, David Piccioni, M.D., Ph.D, Assistant Clinical Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130418
Record Dates: First submitted 2014-01-15; First posted 2014-01-28 (Estimated); Results first posted 2016-08-09 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-08

CONDITIONS: Brain Cancer
Keywords: Brain; Metastasis; human epidermal receptor (HER)
MeSH Terms: conditions — Brain Neoplasms; Neoplasm Metastasis | interventions — dacomitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dacomitinib (Experimental): Dacomitinib 45 mg will be administered orally daily. Treatment cycles will consist of 28 days.
  Interventions: Drug: Dacomitinib

INTERVENTIONS:
Drug: Dacomitinib — Dacomitinib 45 mg will be administered orally daily. Treatment cycles will consist of 28 days.

SUMMARY:
The purpose of this study is to determine the disease response, survival, and side effects of an experimental drug called dacomitinib in progressive brain metastases.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the use of the irreversible pan-ErB kinase inhibitor dacomitinib in the treatment of brain metastases, as measured by radiographic objective response rate.

The rationale of this study is three-fold. First, the use of dacomitinib, an irreversible pan-ErB kinase inhibitor, is to improve the duration of response seen by reversible, EGFR only inhibitors. Inhibition of the multiple ErB kinases may interfere with receptor cross-talk as a method of developing resistance; indeed, patients who have failed erlotinib treatment for systemic disease have seen responses to dacomitinib. The second rationale is to evaluate the pharmacokinetics of the penetration of dacomitinib into the CSF to determine if adequate drug levels reach the CNS, and determine if the current dosing regimen is appropriate. The third rationale is to determine if specific molecular phenotypes preferentially respond to dacomitinib. As part of this study, serum and cerebrospinal fluid will be collected and analyzed both for drug levels and for molecular markers to key elements of the ErB signaling cascade. The objective of the marker analysis to identify a distinct molecular phenotype that may preferentially respond to targeted drug therapy in the future.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) documented extracranial diagnosis of primary lung cancer, melanoma, human epidermal growth factor receptor 2 (HER2)-amplified breast cancer, or HER2-amplified gastric cancer, with brain metastasis detected by contrast enhanced MRI or CT is required. Patients with concurrent leptomeningeal diseases are eligible.
* Has progression and measureable brain disease in the brain by magnetic resonance imaging (MRI) or computed tomography (CT).
* Has stable, or no evidence of, extracranial disease and not receiving systemic therapy for extracranial disease.

Note: Patients with stable disease must have already received standard therapy or are intolerant to standard therapy.

* Prior therapy for brain metastasis is not required; patients may either have refused radiation therapy or have received prior radiation therapy. Patients having received prior standard whole brain radiation therapy (WBRT) or stereotactic radiosurgery (SRS) must have completed treatment greater than 4 weeks prior to study initiation.
* Has recovered from the toxic effects of prior therapy to Common Toxicity Criteria for Adverse Effects (CTCAE) Grade 1 or to their clinical baseline.
* Age ≥18.
* Life expectancy > 3 months in the opinion of the investigator.
* KPS ≥ 60%.
* Adequate organ and marrow function.

Exclusion Criteria:

* Current or planned use of systemic therapy for extracranial primary tumor.
* Current or anticipated use of other investigational agents.
* Presence of uncontrolled seizures ≤ 5 days prior first drug dose, defined as status epilepticus or multiple seizures not responding to appropriate therapy.
* Current or anticipated use of enzyme-inducing anti-epileptic drugs
* Insufficient time for recovery from prior therapy: less than 28 days from WBRT or SRS; less than 28 days from any investigational agent; less than 28 days from prior cytotoxic therapy (except 23 days from prior temozolomide, 14 days from vincristine, 42 days from nitrosoureas, 21 days from procarbazine administration), and less than 7 days for non-cytotoxic agents, e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, etc. When radiation necrosis is suspected, confirmatory imaging will be performed, and patients with findings consistent with radiation necrosis will be excluded.
* Current use or anticipated need for treatment with Coumadin® or other agents containing warfarin (except low dose Coumadin (1 mg or less daily) administered prophylactically for maintenance of in-dwelling lines or ports). Heparin, low molecular weight heparin (LWMH), direct thrombin inhibitors and factor Xa inhibitors are allowed. Rivaroxaban should be used with caution. Antiplatelet agents are allowed.
* Current or anticipated need for treatment with drugs that are known substrates of CYP2D6
* Current or anticipated need for treatment with proton pump inhibitors. Patients on proton pump inhibitors who can be switched to H2-blockers before the start of the study are still eligible.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to dacomitinib.
* Known severe and/or uncontrolled medical disorder that would impair ability to receive study treatment (i.e., uncontrolled diabetes, chronic renal disease, chronic pulmonary disease, HIV, hepatitis B virus (HBV), hepatitis C virus (HCV), or active infection).
* Impaired cardiac function including any of the following: Congenital long QT syndrome or a known family history of long QT syndrome; corrected QT interval (QTc) > 450 msec; history or presence of clinically significant ventricular or atrial tachyarrhythmias; clinically significant resting bradycardia (< 50 beats per minute); myocardial infarction within 1 year of starting study drug; other clinically significant heart disease (e.g., unstable angina, congestive heart failure, or uncontrolled hypertension)
* Pregnant or nursing. There is a potential for congenital abnormalities and for this regimen to harm nursing infants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Piccioni, M.D., Ph.D., Principal Investigator — University of California Medical Center
Locations (1):
- UCSD Moores Cancer Center, La Jolla, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dacomitinib
Started | 4
Completed | 1
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Dacomitinib
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Intra-cranial Objective Response Rate
Description: Intra-cranial objective response rate at 2 months as assessed by the Response Assessment in Neuro-oncology (RANO) criteria
Time Frame: 2 months
Population: Subjects did not complete the study as planned. Zero participants analyzed due to termination of study. Data not available.
Arm/Group | Dacomitinib
Number analyzed (Participants) | 0

2. Secondary Outcome: Treatment-emergent Adverse Events
Time Frame: End of Treatment (4-6 weeks after permanent discontinuation of study treatment for any reason)
Population: The study was terminated due to slow enrollment. Please see adverse event section for additional information.
Arm/Group | Dacomitinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Dacomitinib
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dacomitinib (N=4)
diplopia (Eye disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 2 (2)
nausea/vomitting (Gastrointestinal disorders) | 1 (1)
dry mouth (Gastrointestinal disorders) | 1 (1)
heartburn (Gastrointestinal disorders) | 1 (1)
fatigue (General disorders) | 1 (1)
anemia (Blood and lymphatic system disorders) | 1 (1)
elevated ALT (Blood and lymphatic system disorders) | 1 (1)
elevated AST (Blood and lymphatic system disorders) | 1 (1)
sinusitis (Infections and infestations) | 1 (1)
cough (Infections and infestations) | 1 (1)
thrush (Infections and infestations) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 1 (1)
hyponatremia (Metabolism and nutrition disorders) | 1 (1)
jaw trismus (Musculoskeletal and connective tissue disorders) | 1 (1)
increased creatinine (Renal and urinary disorders) | 1 (2)
rash (Skin and subcutaneous tissue disorders) | 1 (2)
dry skin/cracking (fingertips/nail bed) (Skin and subcutaneous tissue disorders) | 1 (1)
acne (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes